CLINICAL TRIAL: NCT07373314
Title: A Randomized Controlled Trial Comparing Modified Tumescent vs. Conventional Laparoscopic TAPP for Inguinal Hernia Repair
Brief Title: Modified vs. Conventional Laparoscopic TAPP for Inguinal Hernia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Taseen Imran, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exp132
Record Dates: First submitted 2026-01-13; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Inguinal Hernia Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Tumescent Laparoscopic TAPP (MT-TAPP) (Experimental)
  Interventions: Other: Modified Tumescent Laparoscopic TAPP (MT-TAPP) for the first group.
- Conventional Laparoscopic TAPP (CL-TAPP) (Active Comparator)
  Interventions: Other: Conventional Laparoscopic TAPP (CL-TAPP)

INTERVENTIONS:
Other: Modified Tumescent Laparoscopic TAPP (MT-TAPP) for the first group. — In this intervention, participants will undergo laparoscopic inguinal hernia repair using the modified tumescent technique. This technique involves pre-peritoneal infiltration of a solution containing lidocaine, epinephrine, and saline. The tumescent solution is injected into the peritoneum to create a "tumescent" effect, making the tissues easier to dissect and reducing bleeding. This approach aims to improve surgical visibility, reduce operative time, minimize postoperative pain, and shorten the learning curve for less experienced surgeons. The rest of the procedure follows the standard laparoscopic TAPP repair, with mesh placement and peritoneal closure.
  Arms: Modified Tumescent Laparoscopic TAPP (MT-TAPP)
Other: Conventional Laparoscopic TAPP (CL-TAPP) — In this intervention, participants will undergo the conventional laparoscopic transabdominal preperitoneal (TAPP) hernia repair. This standard technique involves placing three ports to access the inguinal region, followed by dissection of the pre-peritoneal space and placement of a mesh to repair the hernia. The conventional method does not use tumescent infiltration and relies solely on the surgeon's skill to navigate the anatomical structures. This approach is well-established and commonly used in inguinal hernia repairs, but it may be associated with longer operative times and more postoperative pain compared to the modified technique.
  Arms: Conventional Laparoscopic TAPP (CL-TAPP)

SUMMARY:
This study aims to compare the outcomes of two laparoscopic techniques for repairing inguinal hernias: the modified tumescent technique (MT-TAPP) and the conventional laparoscopic transabdominal preperitoneal technique (CL-TAPP). The primary goal is to determine which technique provides better outcomes in terms of operative time, ease of pre-peritoneal space dissection, postoperative pain, and the formation of seromas. The study will involve 60 patients diagnosed with unilateral inguinal hernias, randomly assigned to either group. Participants in Group A will undergo the MT-TAPP procedure, which involves pre-peritoneal infiltration of a local anesthetic solution to improve dissection and reduce pain. Group B will undergo the standard CL-TAPP procedure. Data will be collected on various outcome measures and analyzed to identify which technique leads to quicker recovery, less postoperative pain, and fewer complications. The results of this study will help guide surgical decisions and improve patient outcomes in inguinal hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 50 years.
* Gender: Both male and female participants.
* Condition: Diagnosed with unilateral inguinal hernia (as per operational definition).
* Health Status: ASA I-III (American Society of Anesthesiologists physical status classification), indicating that the patient is fit for surgery.
* Consent: Participants must be able to provide informed consent to participate in the study.

Exclusion Criteria:

* Femoral Hernias.
* Incarcerated or Strangulated Hernia.
* Recurrent Hernias (as per medical record).
* Serious Systemic Diseases:
* Conditions such as heart failure or coagulation problems (e.g., PT > 15 sec).
* ASA III-V classification, indicating a higher risk for surgery.
* Pregnancy (if applicable).
* Allergy to Anesthesia or the substances used in the tumescent solution (lidocaine, epinephrine, saline).
* Uncontrolled Diabetes or other medical conditions that might interfere with the healing process.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Pain Score | Recorded 24 hours post-surgery.
  A score of 0 represents no pain, while a score of 10 represents the worst pain.
Seroma Formation: | Presence or absence of seroma, assessed during the 7-day postoperative follow-up.

IPD SHARING:
Plan to Share IPD: No